CLINICAL TRIAL: NCT01007409
Title: Randomized, Open-labeled, Single Dosing Study to Assess Food Effect on the Pharmacokinetics of Fimasartan in Healthy Male Volunteers
Brief Title: A Study to Assess Food Effect on the Pharmacokinetics of Fimasartan in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Choi, Director, Boryung
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: A657-BR-CT-111
Record Dates: First submitted 2009-11-02; First posted 2009-11-04 (Estimated); Last update posted 2009-12-24 (Estimated); Status verified 2009-12

CONDITIONS: Healthy
Keywords: To assess food effect on the pharmacokinetics of fimasartan in healthy male volunteers
MeSH Terms: interventions — fimasartan

ARMS (2):
- Group B (Active Comparator): Period 1: fed control → Period 2: fasted control
  Interventions: Drug: Fimasartan
- Group A (Active Comparator): Period 1: fasted control → Period 2: fed control
  Interventions: Drug: Fimasartan

INTERVENTIONS:
Drug: Fimasartan — Period 1: administration of fimasartan 240mg at 9:00am, 30 minutes after the breakfast Period 2: administration of fimasartan 240mg at 9:00am, without the breakfast
  Arms: Group B
Drug: Fimasartan — Period 1: administration of fimasartan 240mg at 9:00am, without the breakfast Period 2: administration of fimasartan 240mg at 9:00am, 30 minutes after the breakfast
  Arms: Group A

SUMMARY:
To assess food effect on the pharmacokinetics of fimasartan in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* age: 20 - 45 years
* sex: male
* body weight: greater than 55 kg
* written informed consent

Exclusion Criteria:

* known allergy to Fimasartan
* existing cardiac or hematological diseases
* existing hepatic and renal diseases
* existing gastrointestinal diseases
* acute or chronic diseases which could affect drug absorption or metabolism history of any serious psychological disorder
* abnormal diet which could affect drug absorption or metabolism
* positive drug or alcohol screening
* smokers of 10 or more cigarettes per day
* participation in a clinical trial during the last 60 days prior to the start of the study

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-10; Primary Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Cmax, Tmax, AUC, T1/2, CL/F etc. | 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours